CLINICAL TRIAL: NCT05123261
Title: Effects of Mindfulness Based Elder Care (MBEC) on Psychological and Spiritual Well Being of Institutional Seniors With Disability
Brief Title: Effects of Mindfulness Based Elder Care (MBEC) on Psychological and Spiritual Well Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, The Office of Research and Development, Mackay Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MOST-103-2314-B-715-002-MY3
Record Dates: First submitted 2021-04-07; First posted 2021-11-17 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Mental Health Issue
Keywords: long term care institutions; seniors with disability; mindfulness-based elder care; spiritual well-being
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the mindfulness-based elder care (MBEC) therapy (Experimental): The experimental group was offered eight 50-minute courses once a week.
  Interventions: Behavioral: the mindfulness-based elder care (MBEC) therapy
- the routine activities (No Intervention): The control group maintained routine activities. And each CG participant had a weekly visit from the research team.

INTERVENTIONS:
Behavioral: the mindfulness-based elder care (MBEC) therapy — According to the mindfulness-based elder care (MBEC) therapy developed by McBee (2008), the experimental group was offered eight 50-minute courses once a week.
  Arms: the mindfulness-based elder care (MBEC) therapy

SUMMARY:
This study aims to verify the effectiveness of the mindfulness-based elder care (MBEC) therapy developed by McBee (2008) in improving the psychological and spiritual well-being of seniors with disabilities living in residential long-term care institutions in Taiwan.

DETAILED DESCRIPTION:
Background: Existing literature indicates that seniors with disabilities living in long-term care institutions are confronted with such issues as changes in their living environment, institutionalized living schedules, and reduced social interaction, which may affect their mental health and cause spiritual disturbances. In recent years, mindfulness therapy has been increasingly proven to effectively improve individuals' mental health and spiritual well-being. However, the effectiveness of the therapy for seniors with disabilities admitted to residential institutions needs to be further verified by empirical studies.

Purpose: This study aims to verify the effectiveness of the mindfulness-based elder care (MBEC) therapy developed by McBee (2008) in improving the psychological and spiritual well-being of seniors with disabilities living in residential long-term care institutions in Taiwan.

Methods: A Randomized control trial was used. The subjects enrolled in this study were the seniors with disability in the residential long-term care institutions in the northern and central part of Taiwan. The inclusion criteria were the seniors with disabilities who (1) lived in a care institution for over 3 months; (2) were aged 65 years or above; (3) failed to obtain a full score for Barthel Index; (4) were able to communicate in Mandarin or Taiwanese; and (5) had no history of mental illness. According to the intervention scheme, the experimental group was offered eight 50-minute courses once a week, while the control group maintained routine activities. In terms of the evaluation of intervention effectiveness, basic data collection tables, and the Barthel Index were used to collect the information of the included seniors with disabilities on basic demography, and ability to perform daily activities. The Geriatric Depression Scale-Short-Short Form (GDS-SF), State Trait Anxiety Inventory (STAI), and Spiritual Well-Being Scale (SWBS) were also adopted to understand the included seniors with disabilities depression, anxiety, and spiritual well-being. The data were collected four times: before the intervention, in the middle of the intervention (the fourth week), at the end of the intervention (the eighth week), and the follow-up four weeks after the intervention (the twelfth week). The collected data was analyzed by SPSS 22.0. Descriptive statistics and the independent samples t-test were used to identify the homogeneity of the two groups, and the linear mixed model was used to compare the improvement results of the experimental group alone and the two groups at different time points.

ELIGIBILITY:
* The inclusion criteria were the seniors with disabilities who (1) lived in a care institution for over 3 months; (2) were aged 65 years or above; (3) failed to obtain a full score for Barthel Index; (4) were able to communicate in Mandarin or Taiwanese; and (5) had no history of mental illness.
* The exclusive criteria were residents have the diagnosis of psychotic disorders, infectious diseases, or been hospitalized.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Change in depression summary scores before intervention to 4-week post intervention. | The data were collected before the intervention to week 12: baseline, in the middle of the intervention (the fourth week), at the end of the intervention (the eighth week), and the follow-up four weeks after the intervention (the twelfth week).
  Depression was measured using the Chinese version of the Geriatric Depression Scale-Short-Short Form (GDS-SF). The Geriatric Depression Scale-Short-Short Form scores range from 0 to 15. Higher scores represent an increased level of depressive symptoms and a cut-off value of 5 is commonly indicative of depression.
Change in Anxiety summary scores before intervention to 4-week post intervention. | The data were collected before the intervention to week 12: baseline, in the middle of the intervention (the fourth week), at the end of the intervention (the eighth week), and the follow-up four weeks after the intervention (the twelfth week).
  Anxiety was measured using the Chinese version of the State Trait Anxiety Inventory (STAI). The State Trait Anxiety Inventory measures two types of anxiety - state anxiety, or anxiety about an event. The total scores range from 40-160 and higher scores are positively correlated with higher levels of anxiety.
Change in Spiritual well-being summary scores before intervention to 4-week post intervention. | The data were collected before the intervention to week 12: baseline, in the middle of the intervention (the fourth week), at the end of the intervention (the eighth week), and the follow-up four weeks after the intervention (the twelfth week).
  Spiritual well-being was measured using the Chinese version of the Spiritual Well-Being Scale (SWBS). The Spiritual Well-Being Scale scores range from 20 to 120. Higher scores represent an increased level of spiritual well-being.

SECONDARY OUTCOMES:
Change in Meaning in life summary scores before intervention to 4-week post intervention. | The data were collected before the intervention to week 12: baseline, in the middle of the intervention (the fourth week), at the end of the intervention (the eighth week), and the follow-up four weeks after the intervention (the twelfth week).
  Meaning in life was measured using the Purpose in Life Test (PIL). The Purpose in Life Test scores range from 20-140 and higher scores are represent an higher level of meaning and purpose in respondents' lives.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Heng Chen, PhD, Principal Investigator — Department of Nursing, Mackay Medical College
Locations (1):
- Department of Nursing, New Taipei City, Taiwan

REFERENCES:
- [Derived] Hsiung Y, Chen YH, Lin LC, Wang YH. Effects of Mindfulness-Based Elder Care (MBEC) on symptoms of depression and anxiety and spiritual well-being of institutionalized seniors with disabilities: a randomized controlled trial. BMC Geriatr. 2023 Aug 18;23(1):497. doi: 10.1186/s12877-023-04220-6. PMID 37596549